CLINICAL TRIAL: NCT01928303
Title: Predicting Oxycodone Dose From Oral Fluid Drug Levels For Chronic Pain Management Patients
Brief Title: Predicting Oxycodone Dose From Oral Fluid Drug Levels
Acronym: AFTSLabs
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Neel Mehta, Assistant Attending of Anesthesiology, Weill Medical College of Cornell University
Other Study IDs: 1212013319
Record Dates: First submitted 2013-08-16; First posted 2013-08-23 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Pain
Keywords: opioids; chronic pain; oxycodone; oxymorphone; patients using opioid pain medication
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Once received into the laboratory at AFTS labs, oral fluid, blood and urine specimens will be aliquoted for analysis, and any remaining sample will be transferred to long term storage at -20 - 0°C.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Pain Patients taking opioid medications: Oral fluid, blood and urine samples will be obtained from chronic pain patients who are taking pain medications from the opioid class of drugs.
- Negative controls: At least 10% of the total subject population. Chronic pain patients who are not taking pain medication from the opioid class of drugs.

SUMMARY:
This study will develop and test an algorithm that will estimate drug dosage from drug levels measured in oral fluid (saliva). Traditionally, urine has been used as the principle medium to monitor drug compliance in patients receiving opioids for chronic pain as well as those being treated for substance abuse. Recently, the use of saliva as an alternative to urine drug testing has been gaining in popularity. Oral fluid has several advantages over urine as a medium for drug screening. In this study, oral fluid, urine and blood specimens will be collected from volunteer patient donors with chronic pain taking opioid medications. Samples from the anonymous donor will be analyzed for opiate class drugs, using New York State Department of Health approved and validated laboratory methods. Analytical results and other information collected will assist in evaluating the use of oral fluid as a specimen to detect opiate drug levels. The measurement of drug concentrations in blood and oral fluid simultaneously will allow for the determination of the amount of oral fluid that will be needed for successful drug testing. It is proposed that by measuring oral fluid drug levels an estimate of the amount of drug taken will be possible.

DETAILED DESCRIPTION:
Each potential subject will be requested to verify their willingness to participate in the study by signing and dating an Informed Consent Form and the Health Insurance Portability and Accountability Act (HIPAA) Authorization for use of protected health information in research.

The donor will produce a sample by placing a collection swab under his or her tongue until the indicator window turns blue. To ensure the validity of the sample, the donor may not eat, drink, or consume candy for ten minutes prior to the collection time.

A second oral fluid sample will be obtained for the purpose of determining salivary pH at the time of collection. The donors will expel oral fluid into a small collection cup or spoon, and the collector will determine pH using specialized pH strips.

Urine samples will be collected from donors in approved specimen cups according to protocols indicated by the New York State Department of Health guidelines. Blood samples will be collected by trained and certified medical professionals using appropriate collection tubes.

Participating donors will also be requested to complete a questionnaire regarding information including age, weight, and medication information (including type of medication, dosage, dosing pattern, and time of last dose), and medical history (concerning known health issues).

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 72 years of age
* Chronic pain patient at Weill Cornell Medical College Pain Medicine Center

Exclusion Criteria:

* taking any medications that can alter the metabolism of oxycodone or oxymorphone in the body
* not a chronic pain patient at Weill Cornell Medical College Pain Medicine Center

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be generally healthy males and females who are undergoing treatment for chronic pain.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
original dose of drug consumed (mg) as predicted by the drug concentration in the oral fluid (ng/mL) | subjects will be followed for 6 months after enrollment.
  The primary goal of the study is to develop and test an algorithm that will estimate drug dosage from measured oral fluid drug levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College Pain Medicine Center, New York, New York, United States

REFERENCES:
- [Background] Bush DM. The U.S. Mandatory Guidelines for Federal Workplace Drug Testing Programs: current status and future considerations. Forensic Sci Int. 2008 Jan 30;174(2-3):111-9. doi: 10.1016/j.forsciint.2007.03.008. Epub 2007 Apr 16. PMID 17434274
- [Background] Cone EJ, Clarke J, Tsanaclis L. Prevalence and disposition of drugs of abuse and opioid treatment drugs in oral fluid. J Anal Toxicol. 2007 Oct;31(8):424-33. doi: 10.1093/jat/31.8.424. PMID 17988455
- [Background] Cone EJ, Presley L, Lehrer M, Seiter W, Smith M, Kardos KW, Fritch D, Salamone S, Niedbala RS. Oral fluid testing for drugs of abuse: positive prevalence rates by Intercept immunoassay screening and GC-MS-MS confirmation and suggested cutoff concentrations. J Anal Toxicol. 2002 Nov-Dec;26(8):541-6. doi: 10.1093/jat/26.8.541. PMID 12501910
- [Background] Crouch D, Day J, Baudys J. Evaluation of aliva/oral fluid as an alternate drug testing specimen. NIJ Report 605-04 (2004).
- [Background] Heit HA, Gourlay DL. Urine drug testing in pain medicine. J Pain Symptom Manage. 2004 Mar;27(3):260-7. doi: 10.1016/j.jpainsymman.2003.07.008. PMID 15010104
- [Background] Hemeryck A, Belpaire FM. Selective serotonin reuptake inhibitors and cytochrome P-450 mediated drug-drug interactions: an update. Curr Drug Metab. 2002 Feb;3(1):13-37. doi: 10.2174/1389200023338017. PMID 11876575
- [Background] Jickells, S and Negrusz, A (editors). (2008) Clarke's Analytical Forensic Toxicology. London: Pharmaceutical Press
- [Background] Lacy, C, Armstrong, L, Golman, M, and Lance, L (editors). (2011) Drug Information Handbook (20th ed). Hudson, OH: Lexicomp
- [Background] Speckl IM, Hallbach J, Guder WG, Meyer LV, Zilker T. Opiate detection in saliva and urine--a prospective comparison by gas chromatography-mass spectrometry. J Toxicol Clin Toxicol. 1999;37(4):441-5. doi: 10.1081/clt-100102434. PMID 10465240